CLINICAL TRIAL: NCT04359173
Title: A Retrospective Propensity Score Matched Analysis Reveals Superiority of Hypothermic Machine Perfusion Over Static Cold Storage in Deceased Donor Kidney Transplantation.
Brief Title: Propensity Score Matched Comparison of HMP vs. SCS in Kidney Transplantation
Acronym: HMP
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: HMP_SCS
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Delayed Graft Function
Keywords: kidney transplantation
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothermic machine perfusion (HMP): patients who underwent kidney transplantation following HMP
- Static cold storage (SCS): patients who underwent kidney transplantation following SCS

SUMMARY:
Hypothermic machine perfusion (HMP) is considered superior to static cold storage (SCS) in kidney transplantation, but the true benefit in the real-world experience remains incompletely understood.

The aim of our study is to investigate the real-world impact of HMP on kidney graft function after deceased donor kidney transplant in an HMP cohort propensity score matched with SCS.

Propensity score matching will be based on CIT, ECD, gender mismatch, CMV mismatch, re-TX and ET-senior program with a caliper of 0.05

ELIGIBILITY:
Inclusion Criteria:

* single kidney transplantation from a deceased donor at Medical University of Innsbruck between 08/2015 and 12/2019

Exclusion Criteria:

* combined kidney transplantation with an other organ
* living donor kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All deceased donor kidney transplants performed between 08/2015 and 12/2019
Sampling Method: Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Delayed graft function (DGF) | 7 days post transplant
  DGF was defined as the need for at least one dialysis within the first seven days after transplant with the exception of dialysis for hyperkalemia or hypervolemia within the first 12 hours post-transplant

SECONDARY OUTCOMES:
graft survival | 24 months post transplant
  24 month graft survival

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schneeberger, Prof., Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No